CLINICAL TRIAL: NCT05773222
Title: The efficAcy and Safety of aPixaban In REal-world Practice in Korean Frail Patients With Atrial Fibrillation: a Prospective Multicenter Non-interventional, Observational Study: ASPIRE Study
Brief Title: Efficacy and Safety of Apixaban in Korean Frail Atrial Fibrillation Patient
Status: Active, not recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eue-Keun Choi, professor, Seoul National University Hospital
Other Study IDs: ASPIRE study
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — apixaban

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Apixaban — Single Group Assignment

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia, and its prevalence is increasing with the aging population [1]. As the prevalence of AF is significantly rising among the population over 70-80 years old and considering the population is at high risk of AF complications such as stroke, oral anticoagulation (OAC) therapy is necessary among these subjects [1-3]. OAC decreases the risk of stroke and systemic thromboembolism with improved mortality among AF patients. The introduction of non-vitamin K antagonist oral anticoagulants (NOAC) has led to more effective and safe anticoagulation therapy among Asian patients [4,5]. Among different types of NOAC, the prescription of apixaban has been increasing based on robust safety data. The ARISTOTLE (Apixaban for Reduction in Stroke and Other Thromboembolic Events in Atrial Fibrillation), phase three clinical trial on apixaban., showed efficacy and safety of apixaban compared to warfarin among 18,000 patients worldwide [6]. However, this study only included 5.5% (986) Asian patients.

Of patients requiring OAC, those of old age, low body weight, or decreased renal function are at 'high risk' of stroke, systemic thromboembolism, and major bleeding events [4, 7-9]. In Korea, among patients prescribed with NOAC due to AF, 35-40% were older than the age of 75 years old, 35% had bodyweight ≤ 60kg and 25-30% had decreased renal function (Creatinine clearance ≤ 60ml/min) [10]. Although apixaban has proved safe in old age, low bodyweight decreased renal function in ARISTOTLE subgroup analyses, the efficacy and safety data on Asian AF patients with high-risk factors is limited [11-14].

In this study, the investigators aimed to evaluate the efficacy and safety of apixaban among high-risk Korean patients in old age, low bodyweight or decreased renal function using a multicenter observational study design

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be ≥19 years.
2. Patient has non-valvular atrial fibrillation necessitating the use of apixaban for stroke prevention.
3. Subjects satisfies single dose reduction criterion for apixaban; (1) age 80 years or older (2) body weight 60kg or lower (3) serum creatinine 1.5mg/dL or higher.

Exclusion Criteria:

1. Patient is vulnerable (according to Korean Good Clinical Practice definition) or disagree with the study.
2. Patient had a history of clinical events, defined as primary and secondary outcomes of the study, prior to study registration after taking apixaban.
3. Patient satisfies two or more dose reduction criteria for apixaban.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A. Arm Label: prospective, multicenter, non-interventional observational study B. Arm type: no intervention
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2019-08-12 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Stroke | up to 12 months
Systemic embolism | up to 12 months
Major bleeding | up to 12 months
  ISTH criteria

SECONDARY OUTCOMES:
Death from any cause | up to 12 months
Myocardial infarction | up to 12 months
Composite of major bleeding and clinically relevant nonmajor bleeding | up to 12 months
  ISTH criteria
Any bleeding | up to 12 months
Other adverse events including liver or kidney function abnormalities | up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National university Hostpital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided